CLINICAL TRIAL: NCT06459908
Title: Effects of Robotic Glove Hand Training on Fine and Gross Motor Function and Activities of Daily Living in Patients After Median Nerve Transfer
Brief Title: Effects of Robotic Glove Hand Training in Patients After Median Nerve Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/02103
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Median Nerve Injury
Keywords: Hand Rehabilitation; Nerve transfer Rehabilitation; Robotic Glove

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted group (RG) (Experimental): Patients in group A will perform these exercises while Wearing robotic hand-training gloves. Group A will perform hand exercises with the help of robotic glove assistance for 3 times per day/ 4 times per week, 45 minutes per session for 6 consecutive weeks, Number of total sessions will be 72 .
  Interventions: Other: Robot Glove Hand Training; Other: Conventional Hand Rehabilitation Exercises
- conventional hand rehabilitation exercises (Active Comparator): The control group will receive the same treatment as Robot Assisted group but without any robot-assisted device.Group B will perform hand exercises without the help of robotic glove for 3 times per day/ 4 times per week, 45 minute session for 6 consecutive weeks.Number of total sessions will be 72 .
  Interventions: Other: Conventional Hand Rehabilitation Exercises

INTERVENTIONS:
Other: Robot Glove Hand Training — Robot Assisted group will perform hand exercises with the help of robotic glove assistance for 3 times per day/ 4 times per week, 45 minutes per session for 6 consecutive weeks. Total Number of Sessions will be 72 Hours.
  Arms: Robot-assisted group (RG)
Other: Conventional Hand Rehabilitation Exercises — Conventional therapy group will perform hand exercises without the help of robotic gloves 3 times per day/ 4 times per week, 45 minute session for 6 consecutive weeks.Total number of sessions will be 72.

SUMMARY:
Selective nerve transfers provide an opportunity for restoring the motor function after nerve injuries. Upper-limb robot-assisted therapy has been established as a safe and feasible treatment to complement rehabilitation after neurological injury. The aim of this study is to explore the combined effects of Hand Training with Robotic Glove on fine and gross motor function and activities of daily living in patients after median nerve transfer. The study will be randomized controlled trial. Participants will be recruited through non probability convenience sampling technique. After screening for eligibility, participants will be randomly assigned by balanced pre-randomization into two groups either to a robot-assisted group (RG), participants of this group receiving robot-assisted Hand Rehabilitation with the Syrebo Robotic Gloves or to a control group (CG), receiving dose-matched conventional Hand Rehabilitation without the robot. Participants will be engaged in exercises 4 times a week for 6 weeks, each participants will receive 3 Hand Rehabilitation therapy sessions of 45 Mins per day focusing on hand function. Data will be assessed at the start of the 1st session and at the end of the last session after 6 weeks with the help of Sollerman Hand Function test, Jebsen Taylor Hand Function test, The Original Barthel Index for Activities of Daily living. Data will be analyzed using SPSS version 25

DETAILED DESCRIPTION:
Selective nerve transfers provide an opportunity for restoring the motor function after nerve injuries. Over the past decade different hand rehabilitation protocols and exercises are developed, robotic assisted rehabilitation is one of them. Upper-limb robot-assisted therapy has been established as a safe and feasible treatment to complement rehabilitation after neurological injury. Robots can precisely control the interaction with the user (e.g., supporting or resisting in an assist-as-needed manner) and render virtual environments both visually and mechanically, making them ideal tools for sensorimotor training, providing engaging and challenging therapy. The aim of this study is to explore the combined effects of Hand Training with Robotic Glove on fine and gross motor function and activities of daily living in patients after median nerve transfer. The study will be randomized controlled trial. Participants will be recruited through non probability convenience sampling technique. After screening for eligibility, participants will be randomly assigned by balanced pre-randomization into two groups either to a robot-assisted group (RG), participants of this group receiving robot-assisted Hand Rehabilitation with Syrebo Robotic Gloves or to a control group (CG), receiving dose-matched conventional Hand Rehabilitation without the robot. The participants will be engaged in exercises 4 times a week for 6 weeks, each participants will receive three Hand Rehabilitation therapy sessions per day focusing on hand function. Each therapy session will be of 45 minutes. These sessions will be embedded in the weekly therapy plan for each individual participant. Data will be assessed at the start of the 1st session and at the end of the last session after 6 weeks with the help of Sollerman Hand Function test, Jebsen Taylor Hand Function test, The Original Barthel Index for Activities of Daily living. Data will be analyzed using SPSS version 25. Key words: Hand Rehabilitation, Nerve transfer Rehabilitation, Robotic Glove

ELIGIBILITY:
Inclusion Criteria:

* Both Genders will be recruited
* Age between 19 to 55 years
* Median nerve transfer after traumatic event (RTA, history of Fall, avulsion, compression or stretch injuries)
* The ability to follow and respond to verbal commands

Exclusion Criteria:

subjects will be excluded if they have

* Altered state of consciousness,
* Aphasia ,
* Severe cognitive deficits .
* Severe pathologies of upper limb of rheumatic nature
* Could not provide informed consent for study
* Severe pain in affected arm Visual analogue scale > 5

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
THE SOLLERMAN HAND FUNCTION TEST (SHT) | 6 Weeks
  Sollerman Hand Function Test (SHT) is an assessment tool for analyzing hand function and grip strength after hand surgery for recording the recovery rate in rehabilitation phase. The scale include 8 hand grips that further divided into 20 subsets that helps in analyzing hand grip pattern that used for daily activities. Further; each activity was scored form 0 to 4 points with collective score of 80. The lower the score the poor hand function and grip strength was observed. SHT considered as most reliable and valid tool in analyzing hand function with excellent inter-rater reliability (ICC:0.987) and moderate test-retest reliability.
JABSEN-TAYLER HAND FUNCTION TEST | 6 Weeks
  Jabsen-Tayler Hand Function Test is an effective assessment tool in analyzing fine and gross motor activity of hand that are required for performing daily activities of life.
  The scale included 7 subsets of activities including writing; turning page, lifting objects; feeding and sacking. It is considered as good to excellent reliable and valid tool with the ICC of 0.77 in dominant hand and 0.84 to 0.97 in non-dominant hand in injured hand.Higher score means worse outcome and Lower score means good outcome.
PEGBOARD TEST | 6 Weeks
  Pegboard Test is a valid instrument that used for assessing hand dexterity movement.Higher score means worse outcome and Lower score means good outcome.
  among the individual. It is a test board having five subsets focusing placing pins, bimanual task performance and mathematical problems. The whole test is scored based on the completion of each subset. It has an excellent validity with ICVI= 0.9-1.0, SCVI = 0.93-0.95 and ICCs =0.76-0.85.
The Original Barthel Index for Activities of Daily Living (ADLs) | 6 Weeks
  The Barthel Index (BI) measures the extent to which somebody can function Independentlybladder control, toileting, chair transfer, ambulation and stair climbing. Items are weighted according to the level of nursing care required and are rated in terms of whether individuals can perform activities independently, with some assistance, or are dependent (scored as 10, 5 or 0). It has 0.89 test-retest reliability and 0.95 internal reliability. Reliability study found an alpha Cronbach value of 0.90 for the complete scale.(30)Higher the score for barthal index it means good outcome and lower the score means poor outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Ghurki Trust Teaching Hospital , Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geuna S, Raimondo S, Ronchi G, Di Scipio F, Tos P, Czaja K, Fornaro M. Chapter 3: Histology of the peripheral nerve and changes occurring during nerve regeneration. Int Rev Neurobiol. 2009;87:27-46. doi: 10.1016/S0074-7742(09)87003-7. PMID 19682632
- [Background] Rydevik B, Lundborg G. Permeability of intraneural microvessels and perineurium following acute, graded experimental nerve compression. Scand J Plast Reconstr Surg. 1977;11(3):179-87. doi: 10.3109/02844317709025516. PMID 609900
- [Background] George SC, Burahee AS, Sanders AD, Power DM. Outcomes of anterior interosseous nerve transfer to restore intrinsic muscle function after high ulnar nerve injury. J Plast Reconstr Aesthet Surg. 2022 Feb;75(2):703-710. doi: 10.1016/j.bjps.2021.09.072. Epub 2021 Oct 22. PMID 34789435
- [Background] Liu Y, Lao J, Gao K, Gu Y, Xin Z. Outcome of nerve transfers for traumatic complete brachial plexus avulsion: results of 28 patients by DASH and NRS questionnaires. J Hand Surg Eur Vol. 2012 Jun;37(5):413-21. doi: 10.1177/1753193411425330. Epub 2011 Nov 8. PMID 22067298
- [Background] Yurkewich A, Kozak IJ, Ivanovic A, Rossos D, Wang RH, Hebert D, Mihailidis A. Myoelectric untethered robotic glove enhances hand function and performance on daily living tasks after stroke. J Rehabil Assist Technol Eng. 2020 Dec 15;7:2055668320964050. doi: 10.1177/2055668320964050. eCollection 2020 Jan-Dec. PMID 33403121